CLINICAL TRIAL: NCT02030470
Title: Evaluation of Photodynamic Treatment FOTOSAN® Efficacy in Periodontology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5716
Record Dates: First submitted 2013-12-16; First posted 2014-01-08 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis
Keywords: Periodontitis, treatment, photodynamic, mid-term, bacteria
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- fotosan (Other)
  Interventions: Other: Fotosan®630. LED lamp. Toluidinblue. Photoactivated disinfection

INTERVENTIONS:
Other: Fotosan®630. LED lamp. Toluidinblue. Photoactivated disinfection

SUMMARY:
Periodontitis are infectious and inflammatory diseases of gum and tooth supporting tissues leading to tooth loss and oral disability. Twenty to 30 percents of patients treated for periodontal diseases display more or less pronounced persistence of periodontal tissue infection, inflammation, and destruction. The therapeutic additional value of photodynamic anti-infectious treatment remains controversial. The objective of this study is to evaluate the mid-term effect of the photodynamic device Fotosan®630 on severe periodontitis treatment outcomes and to define its specific therapeutic indications.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 years
* signed informed consent
* generalized severe chronic periodontitis
* patient with at least 24 teeth
* more than 30% of sites with clinical attachment loss >5mm- at least 5 sites with pocket depth >4mm per quadrant- at least one molar per quadrant- evidenced bone loss on radiographs- bleeding on probing ≥30%

Exclusion Criteria:

* aggressive periodontitis
* smoking more than 10cig/day
* patient with endocarditis risk or need of antibiotic prophylaxis
* pregnant women
* patient included in other trials
* patient under guardianship
* patient treated with antibiotics, anti-inflammatory, and other drugs (inhibitors of calcium channels…) influencing periodontal status within 6 months before examination
* patient suffering from diseases influencing periodontal status (diabetes…)
* patient periodontally treated with root planing or periodontal surgery within 1 year before examination
* patient with scheduled extensive prosthetic treatment
* patient with a high haemorrhagic risk (INR>4)
* impossible patient cooperation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of periodontal pocket depth | 6 months
  Study period for each participant : 6 months Inclusion period: 24 monthTotal study duration: 30 month

SECONDARY OUTCOMES:
Change of periodontal clinical attachment level, gingival inflammation and dental plaque indexChange of periodontal microflora | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Davideau, MDPHD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de parodontologie, Strasbourg, Alsace, France

REFERENCES:
- [Result] Harmouche L, Courval A, Mathieu A, Petit C, Huck O, Severac F, Davideau JL. Impact of tooth-related factors on photodynamic therapy effectiveness during active periodontal therapy: A 6-months split-mouth randomized clinical trial. Photodiagnosis Photodyn Ther. 2019 Sep;27:167-172. doi: 10.1016/j.pdpdt.2019.05.022. Epub 2019 May 19. PMID 31116996
- [Derived] Courval A, Harmouche L, Mathieu A, Petit C, Huck O, Severac F, Davideau JL. Impact of Molar Furcations on Photodynamic Therapy Outcomes: A 6-Month Split-Mouth Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Jun 11;17(11):4162. doi: 10.3390/ijerph17114162. PMID 32545223